CLINICAL TRIAL: NCT04324814
Title: A Phase 1, Open-Label, Multi-Center, Non-Randomized, Dose Escalation/Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of SHR-1701 in Subjects With Advanced Solid Tumors.
Brief Title: A Trial of SHR-1701 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-001AUS
Record Dates: First submitted 2019-11-28; First posted 2020-03-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — SHR-1701

STUDY DESIGN:
Intervention Model Description: Dose escalation is designed according to a modified 3+3 scheme, in which 3 to 6 subjects will be enrolled in each dose group. Four dose levels of SHR-1701 are planned. After completion of dose escalation, selected cohort(s) will be expanded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose level 1 (Experimental): Subjects will receive a single dose of SHR-1701 at Dose level 1 on Day 1 of each cycle
  Interventions: Drug: SHR-1701
- Dose level 2 (Experimental): Subjects will receive a single dose of SHR-1701 at Dose level 2 on Day 1 of each cycle
  Interventions: Drug: SHR-1701
- Dose level 3 (Experimental): Subjects will receive a single dose of SHR-1701 at Dose level 3 on Day 1 of each cycle
  Interventions: Drug: SHR-1701
- Dose level 4 (Experimental): Subjects will receive a single dose of SHR-1701 at Dose level 2 1 on Day 1 and Day 15 of each cycle
  Interventions: Drug: SHR-1701
- Dose level 5 (Experimental): Subjects will receive a single dose of SHR-1701 at Dose level 3 on Day 1 and Day 15 of each cycle
  Interventions: Drug: SHR-1701
- Dose expansion 1 (Experimental): Subjects will receive a single dose of SHR-1701 on a selected dose level Day 1 of each cycle
  Interventions: Drug: SHR-1701
- Dose expansion 2 (Experimental): Subjects will receive a single dose of SHR-1701 on a selected dose level on Day 1 of each cycle
  Interventions: Drug: SHR-1701

INTERVENTIONS:
Drug: SHR-1701 — Anti-PD-L1/TGFβ fusion protein

SUMMARY:
This is a dose-escalation and dose-expansion Phase 1 trial to evaluate the safety and tolerability of SHR-1701 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a two-part, open-label, multicenter, non-randomized, dose escalation, Phase 1 study of repeated doses of SHR-1701 in subjects with advanced solid tumors who have failed current standard anti-tumor therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed (histologically or cytologically) with solid tumors
* ECOG Performance Status of 0 or 1 at both the screening and baseline visits
* Life expectancy ≥12 weeks
* Adequate laboratory parameters
* Willing and able to comply with clinic visits and study-related procedures
* Provide signed informed consent

Exclusion Criteria:

* Known history of hypersensitivity to the study drug
* Prior malignancy active within the previous 2 years
* Any investigational or concurrent cancer therapy
* History of immunodeficiency including seropositivity
* Systemic antibiotics treatment for ≥ 7 days before the first dose
* A known history of allogeneic organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | Screening up to study completion, an average of 1 year
  Number of subjects with adverse events (AEs)
Laboratory results | Screening up to study completion, an average of 1 year
  Number of subjects with laboratory tests findings of potential clinical importance
Vital signs | Screening up to study completion, an average of 1 year
  Incidence of vital sign abnormalities
Electrocardiogram | Screening up to study completion, an average of 1 year
  Number of subjects with clinically significant abnormal ECG QT Interval

SECONDARY OUTCOMES:
Pharmacokinetic - Cmax | Pre-dose, 10min(±2min), 1h(±5min), 2h(±5min), 6h(±10min) Post-dose on Cycle1 Day 1, pre-dose on Day 2, 3, 4, 8, 15
  Maximum observed plasma concentration (Cmax) of SHR-1701
Pharmacokinetic - AUC∞ | Pre-dose, 10min(±2min), 1h(±5min), 2h(±5min), 6h(±10min) Post-dose on Cycle1 Day 1, pre-dose on Day 2, 3, 4, 8, 15
  Area under the concentration-time curve from time 0 to infinity of SHR-1701
Pharmacokinetic - Tmax | Pre-dose, 10min(±2min), 1h(±5min), 2h(±5min), 6h(±10min) Post-dose on Cycle1 Day 1, pre-dose on Day 2, 3, 4, 8, 15
  Time to Cmax of SHR-1701
Pharmacokinetic - CL/F | Pre-dose, 10min(±2min), 1h(±5min), 2h(±5min), 6h(±10min) Post-dose on Cycle1 Day 1, pre-dose on Day 2, 3, 4, 8, 15
  Apparent clearance of SHR-1701
Pharmacokinetic - Vz/F | Pre-dose, 10min(±2min), 1h(±5min), 2h(±5min), 6h(±10min) Post-dose on Cycle1 Day 1, pre-dose on Day 2, 3, 4, 8, 15
  Apparent volume of distribution during terminal phase of SHR-1701
Pharmacokinetic - t1/2 | Pre-dose, 10min(±2min), 1h(±5min), 2h(±5min), 6h(±10min) Post-dose on Cycle1 Day 1, pre-dose on Day 2, 3, 4, 8, 15
  Terminal elimination half-life
Pharmacodynamics- ADA | Pre-dose on Day1 of cycle 2,3,4,5,7,9,13,17
  Anti-drug antibody of PD-L1

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Icon Cancer Care Centre, South Brisbane, New South Wales
  - Scientia Clinical research, Sydney, New South Wales
  - Sydney South West Private, Sydney, New South Wales
  - Linear Clinical Research, Perth, Western Australia